CLINICAL TRIAL: NCT01173796
Title: Ablation of Perimitral Flutter Following Catheter Ablation of Atrial Fibrillation: Impact on Outcomes
Acronym: PROPOSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCAI-PROPOSE
Record Dates: First submitted 2010-06-21; First posted 2010-08-02 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Atrial Fibrillation; Perimitral Flutter
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PMFL ablation (Experimental): Radio-frequency catheter ablation of the mitral isthmus only
  Interventions: Procedure: catheter ablation
- Repeat PVAI and triggers ablation (Experimental): cardioversion and repeat isolation of pulmonary veins (PV) with ablation of additional triggers
  Interventions: Procedure: catheter ablation

INTERVENTIONS:
Procedure: catheter ablation — perimitral flutter ablation by blocking the mitral isthmus
  Arms: PMFL ablation
Procedure: catheter ablation — cardioversion and repeat isolation of pulmonary veins (PV) with ablation of additional triggers
  Arms: Repeat PVAI and triggers ablation

SUMMARY:
This prospective, randomized study aims to compare the impact of ablation of perimitral flutter only versus cardioversion and repeat isolation of pulmonary veins with ablation of additional triggers, on procedure outcome.

DETAILED DESCRIPTION:
Background: In recent years, catheter ablation has been accepted as the treatment-of-choice for drug-refractory atrial fibrillation (AF). It is centered around isolating pulmonary veins (PVs) and its success rate in curing AF is very high (56%-85%) (1). However, despite isolation of this dominant source of triggers, recurrent tachyarrhythmia is the major complication of this procedure with peri-mitral atrial flutter (PMFL) being the most common macro-reentrant arrhythmia in context of AF ablation (2). These often drug-refractory arrhythmias are frequently associated with more severe symptoms than the original AF (3) and warrant the necessity for redo-ablation.

This study aims to compare the impact of two different redo-ablation strategies on the procedure outcome; (1) ablation of the perimitral flutter only and (2) cardioversion and repeat isolation of pulmonary veins (PV) with ablation of additional triggers.

Study method: A total number of 65 AF patients presenting for redo-ablation and PMFL will be randomized to perimitral flutter ablation only or cardioversion and re-isolation (PVI) plus ablation of additional triggers. Additional triggers will be identified with the help of post-ablation drug provocation with isoproterenol. Patients will enter a follow-up period of 12 months after the ablation procedure, when they will be monitored for recurrence of arrhythmia detected either by in-clinic or remote device interrogation at 1, 3, 6 and 12 month post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previous AF ablation presenting with PMFL and recurrent AF
* Age: 18- 75 years
* Willingness and ability to give written informed consent
* Therapeutic INR for at least 4 weeks prior to the procedure

Exclusion Criteria:

* Reversible causes of AF such as pericarditis and hyperthyroidism
* Documented intra-atrial thrombus, tumor or any other abnormality which prevents easy catheter manipulation
* Enrollment in another clinical study
* Any other terminal illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Freedom from AF/ flutter/ tachycardia off antiarrhythmic therapy | 1 year

SECONDARY OUTCOMES:
Total number of hospitalizations during the study period Change in quality of life | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas cardia Arrhythmia Institute, St.David's Medical center
Locations (1):
- Texas Cardiac Arrhythmia Research Foundation, Austin, Texas, United States

REFERENCES:
- [Derived] Bai R, Di Biase L, Mohanty P, Dello Russo A, Casella M, Pelargonio G, Themistoclakis S, Mohanty S, Elayi CS, Sanchez J, Burkhardt JD, Horton R, Gallinghouse GJ, Bailey SM, Bonso A, Beheiry S, Hongo RH, Raviele A, Tondo C, Natale A. Ablation of perimitral flutter following catheter ablation of atrial fibrillation: impact on outcomes from a randomized study (PROPOSE). J Cardiovasc Electrophysiol. 2012 Feb;23(2):137-44. doi: 10.1111/j.1540-8167.2011.02182.x. Epub 2011 Sep 28. PMID 21955215